CLINICAL TRIAL: NCT01906619
Title: Investigation of the Respiratory Physiology of Children With and Without Febrile Seizures During Febrile Illness.
Brief Title: Respiratory Physiology in Children With Febrile Seizures.
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Sana-Klinikum Lichtenberg (Other)
Responsible Party: Principal Investigator, Markus Schuelke, M.D., Prof. Dr. med. / Prinicpal Investigator, Charite University, Berlin, Germany
Other Study IDs: EA2_009_10
Record Dates: First submitted 2013-07-20; First posted 2013-07-24 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Febrile Illness Acute; Seizures, Febrile
Keywords: Febrile Seizure; Respiratory physiology; Respiratory drive; Respiratory alkalosis
MeSH Terms: conditions — Seizures, Febrile; Alkalosis, Respiratory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Febrile illness WITH febrile seizure: The cohort comprises children aged between 3 months and 5 years who had a febrile seizure during the actual febrile disease.
- Febrile illness WITHOUT febrile seizure: The cohort comprises children aged between 3 months and 5 years with a febrile illness who had never a febrile seizure.

SUMMARY:
Febrile seizures occur in 2-5% of the population and are typically limited to children between 3 months and 5 years-of-age. The pathophysiological link between increased body temperature and increased seizure susceptibility is unsolved in humans. In a mouse model it has been shown that young animals had a tendency to hyperventilate thereby causing intra-cerebral hypocapnia / alkalosis and a decrease of their seizure threshold. This effect was not observed in older animals. Redressing the pCO2 (carbon dioxide partial pressure) by breathing carbon dioxide enriched air instantly stopped the seizures.

In this study the investigators want to investigate the respiratory physiology in children with febrile seizures and compare it to children who have fever but did not have febrile seizures.

The investigators hypothesize that in children with febrile seizures the rising body temperature triggers a larger increase of respiratory rate (hyperventilation) and subsequent drop in pCO2 levels.

This study could provide the basic physiological data for an interventional trial to test the efficacy of carbon dioxide inhalation to interrupt febrile seizures.

DETAILED DESCRIPTION:
The aim of the study is the continuous non-invasive monitoring of

* body temperature
* respiratory rate
* transcutaneous pCO2
* heart rate
* pulsoxymetric SaO2 (arterial oxygen saturation) during a febrile illness
* in children without febrile seizures and
* in children who had suffered a febrile seizure during the actual febrile illness.

Children will be recruited from the emergency units of the Charité University Hospital and a large Community Hospital, matched according to age, gender and the cause of their febrile illness and their data will enter final analysis if their body temperature rose at least once to or above 38.0 degree C and changed more than 1.0 degree C during the observational period.

ELIGIBILITY:
Inclusion Criteria:

* Febrile illness with body temperature ≥38.0 degree C
* 50% of study population: never had a febrile seizure
* 50% of study population: simple or complex febrile seizure within one day of investigation
* Change of body temperature of ≥1.0 degree C during the monitoring period
* Provision of written informed consent by the parents or guardians of the child
* Artefact-free simultaneous measurement of respiratory rate, pCO2 (transcutaneous probe), body temperature (rectal probe), and heart rate during change of body temperature of ≥1.0 degree C.

Exclusion Criteria:

* Past history of afebrile seizures
* Past history of neonatal seizures
* Retarded psychomotor development
* Chronic respiratory disease
* Cardiologic disease
* Severe other organ disease
* Permanent medication for chronic disorder
* Therapeutic increase of inspiratory oxygen concentrations during the observational period

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with febrile illness between 3 months and 5 years of age with a body temperature of >38.0 during the monitoring period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change of transcutaneous pCO2 per change of body temperature [mmHg/degree C] | First or second night of febrile illness
  The following parameters are continuously monitored in the sleeping child at night during febrile illness: body temperature, respiratory rate, transcutaneous pCO2, heart rate, pulsoxymetric SaO2
Change of respiratory rate per change of body temperature [1/sec * degree C] | First or second night of febrile illness
  The following parameters are continuously monitored in the sleeping child at night during febrile illness: body temperature, respiratory rate, transcutaneous pCO2, heart rate, pulsoxymetric SaO2
Change of transcutaneous pCO2 per change of respiratory rate [mmHg * sec] | First or second night of febrile illness
  The following parameters are continuously monitored in the sleeping child at night during febrile illness: body temperature, respiratory rate, transcutaneous pCO2, heart rate, pulsoxymetric SaO2

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schuelke, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany